CLINICAL TRIAL: NCT02226887
Title: "Prospective Randomized Clinical Trial of Ileostomy Closure Site Hernia and it´s Prophylaxis by Placing an Absorbable Mesh "
Brief Title: Prophylaxis of Ileostomy Closure Site Hernia by Placing Mesh
Acronym: ILEOCLOSE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PR(AG)288/2013
Record Dates: First submitted 2014-03-18; First posted 2014-08-27 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Loop Ileostomy Closure
Keywords: Loop ileostomy; Eventration
MeSH Terms: conditions — Gastroschisis | interventions — Hematologic Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- MESH (Experimental)
  Interventions: Procedure: MESH; Radiation: Post-operative Imaging; Radiation: Pre-operative Imaging; Other: Blood Test and C-reactive protein at 4th day
- NO MESH (Active Comparator)
  Interventions: Procedure: NO MESH; Radiation: Post-operative Imaging; Radiation: Pre-operative Imaging; Other: Blood Test and C-reactive protein at 4th day

INTERVENTIONS:
Procedure: MESH — 1. Pre-operative :
     It was made by barium enema protocol and transanal endoscopy to rule out anastomotic leaks or strictures contraindicating stoma closure .
  2. Surgical technique:
     * Peristomal incision with electrocautery
     * Release the handle of ileum
     * Anastomosis made the with the segment everted sutured by simple manual end to end 3/0 or mechanical side to side (surgeon's election).
     * Return the ileum into the abdominal cavity and the fascial defect is repaired with continuous polydioxanone 1/0 suture respecting 4:1 measurement rule.
     * We add the mesh between the edges of the defect during fascia closure.
     * The skin is sutured "purse string" style.
  3. Post-Op
     * Hospital discharge after verification of normal digestive transit.
  Other Names: Mesh : GORE® BIO-A®
  Arms: MESH
Procedure: NO MESH — 1. Pre-operative :
     It was made by barium enema protocol and transanal endoscopy to rule out anastomotic leaks or strictures contraindicating stoma closure .
  2. Surgical technique:
     * Peristomal incision with electrocautery
     * Release the handle of ileum
     * Anastomosis made the with the segment everted sutured by simple manual end to end 3/0 or mechanical side to side (surgeon's election).
     * Return the ileum into the abdominal cavity and the fascial defect is repaired with continuous polydioxanone 1/0 suture respecting 4:1 measurement rule.
     * The skin is sutured "purse string" style.
  Post-Op
  - Hospital discharge after verification of normal digestive transit
  Other Names: Protocol Ileostomy closure
  Arms: NO MESH
Radiation: Post-operative Imaging — Abdominal Tomography 1 year after ileostomy closure
Radiation: Pre-operative Imaging — Contrast study is used to ensure the integrity of the distal anastomosis
Other: Blood Test and C-reactive protein at 4th day — All patients undergo a Blood Test study of C-reactive protein on day 4 by protocol within the unit before discharge.

SUMMARY:
Design Prospective , randomized, parallel phase IV.

Objectives Main objective

* Evaluate the effectiveness of the placement of a resorbable mesh in the prevention of incisional hernia of the abdominal wall at the site of a loop ileostomy when it is "closed " to rebuild the intestinal transit. The effectiveness evaluation is done by tracking with scheduled patient visits for 12 months, assessing the physical examination the presence or absence of an incisional hernia and an abdominal tomography at the end of the 12 months .

Secondary objectives Comparison of complications(morbidity and mortality) to assess safety and tolerability of the placement of the mesh described .

DETAILED DESCRIPTION:
Experimental: Reinforcement with Absorbable Mesh Closure of the ileostomy closure incision is reinforced with insertion of a rectangular segment (1 cm wide and the length corresponding to the incision) of a prosthetic commercially available GORE® BIO-A® Tissue Reinforcement prosthesis (W. L. Gore & Associates, Flagstaff, Arizona, USA) mesh. The BIO-A® prosthesis is inserted using a "sandwich" method between the edges of the incision and maintained in situ with a continuous polydioxanone (PDS) suture following a suture length to wound length (SL:WL) ratio of 4:1.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a loop ileostomy closure

Exclusion Criteria:

* Patients under 18
* Pregnancy and Lactation
* Patients allergic to polyglycolic / trimethylene carbonate
* Carrier of prosthetic mesh in the ostomy
* Patients presenting midline hernia.
* Patients affected by inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Eventration | 1 year
  Measured by clinical checks at 1 - 6 - 12 months and Abdominal tomography 1 year after the surgery.

SECONDARY OUTCOMES:
Occlusive problems | 30 days after surgery
  Intestinal occlusion, Anastomotic stenosis, Prolonged ileus(>5days),....
  * This is a Clinical measure supported by image if necessary
  * All the morbidity problems are reported independently.
  * 1 patient can suffer a prolonged ileus and Anastomotic stenosis and both will be reported.
Iatrogenic problems | 30 days after surgery
  Damage to structures such as ureters, bowel loops artery / iliac vein ....
  * This is a Surgical and Clinical measure supported by image if necessary.
  * All the morbidity problems are reported independently.
Impaired healing | 30 days after surgery
  Anastomotic leak rate , intestinal fistula , vesical fistula, peritonitis...
  * This is a Clinical measure always supported by image tests.
  * All the morbidity problems are reported independently.
Bleeding problems | 30 days after surgery
  Hemoperitoneum, abdominal hematoma,anastomotic bleeding ....
  * This is a Clinical measure supported by image if necessary.
  * All the morbidity problems are reported independently.
  * The amount of blood loss won't be specified
Cardiac complications | 30 days after surgery
  acute myocardial infarction, angor pectoris , atrial fibrillation, acute pulmonary edema
  * This is a Clinical measure supported by more specific tests if necessary.
  * All the morbidity problems are reported independently.
  * Cardiologist report will be required for including this items
Nephro-urinary complications | 30 days after surgery
  Acute urinary retention, Acute renal failure, cystitis, pyelonephritis ...
  * This is a Clinical measure supported by more specific tests if necessary.
  * All the morbidity problems are reported independently.
Respiratory complications | 30 days after surgery
  Pneumonia, Atelectasis, Pulmonary embolism, Respiratory distress syndrome ...
  * This is a Clinical measure always supported by image .
  * All the morbidity problems are reported independently.
Vascular Complications | 30 days after surgery
  Deep venous thrombosis, phlebitis, thrombophlebitis, ...
  * This is a Clinical measure supported by more specific test if necessary .
  * All the morbidity problems are reported independently
Gastrointestinal complications | 30 days after surgery
  Liver failure, gastrointestinal bleeding, severe malnutrition, ...
  * This is a Clinical measure supported by blood test and further test if necessary
  * All the morbidity problems are reported independently.
Neurological complications | 30 days after surgery
  Disorientation, cerebral vascular accident, ...
  * This is a Clinical measure.
  * All the morbidity problems are reported independently.
  * Neurologist report will be required beyond disorientation.
Local infection | 30 days after surgery
  Superficial, deep, body-cavity
  * This is a Clinical measure supported by image if necessary
  * All the morbidity problems are reported independently
Local complications | 30 days after surgery
  Hematoma, seroma, evisceration
  * This is a Clinical measure
  * All the morbidity problems are reported independently
Hospital stay | Days
  Hospital stay since surgery is done

CONTACTS AND LOCATIONS:
Overall Officials: Borja Villanueva Figueredo, MD, Principal Investigator — Hospital Universitari Vall d'Hebron Research Institute; Francesc Vallribera Valls, MD,PhD, Study Director — Hospital Universitari Vall d'Hebron Research Institute; Manuel Lopez-Cano, MD, PhD, Study Director — Hospital Universitari Vall d'Hebron Research Institute
Locations (1):
- Hospital General Universitario Vall d´Hebron, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No